CLINICAL TRIAL: NCT06062771
Title: A Prospective, Single-center, Within Patient Randomized, Noninferiority, Controlled, Single-masked Clinical Investigation to Evaluate Efficacy and Safety of the Use of Ophthalmic Viscosurgical Devices (OVD) FIDIAL PLUS vs IAL®-F During Cataract Surgery
Brief Title: Efficacy and Safety of the Use of Ophthalmic Viscosurgical Devices (OVD) FIDIAL PLUS vs IAL®-F During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: QQ24_20_01
Record Dates: First submitted 2023-06-13; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cataract
Keywords: Ophthalmic Viscosurgical Devices; Corneal endothelium cells; Cataract Surgery; Hyaluronic acid
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Each eye will be randomly assigned to Test or Reference such as the subject has one eye treated with FIDIAL PLUS solution and the other with IAL-F solution. For all subjects the worst eye will be operated on first.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIDIAL PLUS (Experimental): Solution of NaHA 20 mg/1.1 ml pre-filled syringe for intraocular use. 1.8% solution of sodium hyaluronate that is derived from a bacterial fermentation (not of animal origin).
  Interventions: Device: FIDIAL PLUS
- IAL®-F (Active Comparator): Solution of NaHA 20 mg/1.1 ml pre-filled syringe for intraocular use. Animal derived 1.8% sodium hyaluronate OVD.
  Interventions: Device: IAL®-F

INTERVENTIONS:
Device: FIDIAL PLUS — 1.8% solution of sodium hyaluronate that is derived from a bacterial fermentation (not of animal origin).
  Arms: FIDIAL PLUS
Device: IAL®-F — Animal derived 1.8% sodium hyaluronate equivalent to FIDIAL PLUS
  Arms: IAL®-F

SUMMARY:
This is a Prospective, single-center, randomized, controlled, paired-eye, single-masked clinical investigation to compare the efficacy and safety of FIDIAL PLUS (bacterial derived 1.8% sodium hyaluronate OVD) and IAL®-F (comparable animal derived 1.8% sodium hyaluronate OVD) while used during phacoemulsification cataract surgery.

DETAILED DESCRIPTION:
Viscoelastics, also referred to as OVDs (ophthalmic viscosurgical devices), are viscous substances that are routinely used in cataract surgery. The most basic benefit of OVD use in ophthalmic surgery is maintaining the anterior chamber during surgical maneuvers. One of the main aspects in OVD use remains the protection of intraocular structures and in particular of corneal endothelium cells (CECs) during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject able to comprehend the full nature and the purpose of the study;
2. Subjects able to cooperate with the Investigator and to comply with the requirements of the entire study;
3. Subject provided written informed consent to participate in the study obtained according to Good Clinical Practice (GCP);
4. Females of childbearing potential (i.e., not permanently sterilised - post hysterectomy or tubal ligation status - or not postmenopausal) must have a negative urine pregnancy test result at Screening and surgery days and must use an appropriate method of contraception for at least 30 days before inclusion in the study and during the whole study period, according to the definition in ICH M3 Guideline.

The following criteria apply to both eyes:

1. Nuclear cataract with visual acuity between 20/200 (logmar 1.0) and 20/32 (logmar 0.2);
2. Intraocular pressure (IOP) between 14 and 21 mmHg (Goldmann tonometer);
3. Previous refraction between -5 and +3 diopters in spherical equivalent;
4. Corneas perfectly transparent without leukoma or other corneal pathology.

Exclusion Criteria:

1. Any acute, chronic or uncontrolled disease as severe heart failure, recent cardiovascular event, respiratory failure, severe hepatic or renal disease, poorly controlled diabetes mellitus, active severe autoimmune disease, active malignancy etc. that in the opinion of the Investigator, would increase the risk of operation or affect the outcome of the study;
2. Epilepsy and any other condition that would prevent cooperation during surgery, including head tremor, deafness, neck or back problems, restless legs syndrome, claustrophobia etc.;
3. Have a history of allergic/hypersensitivity reaction to sodium hyaluronate (NaHA);
4. Participation in another clinical trial within the past 30 days;

The following criteria apply both eyes:

1. Corneal endothelium cell density less than 1800 cells/mm square;
2. Pseudoexfoliation syndrome (PEX) or suspected zonular compromise of any origin;
3. Corneal angle narrow or/and glaucoma;
4. Anterior segment pathology likely to increase the risk of an adverse outcome for phacoemulsification cataract surgery (e.g., pseudoexfoliation syndrome, synechiae, iris atrophy, inadequate dilation, shallow anterior chamber, traumatic cataract, lens subluxation etc.);
5. Any corneal irregularity or leukoma (as assessed by slit lamp and specular microscope pachymetry);
6. Complicated cataracts;
7. Subjects requiring implantation of toric lenses;
8. Proliferative retinopathy, macular degeneration or oedema of any origin. Other ocular pathology that may compromise vision despite successful cataract surgery;
9. Signs of ocular or systemic infection and/or inflammation;
10. Previous intraocular surgery, refractive surgery or severe ocular trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-23 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change of corneal endothelium cell density after phacoemulsification cataract surgery with use of two different OVD (Ophthalmic Viscosurgical Devices) | 28 days per eye
  This outcome will be calculated as percentage of corneal endothelial cells loss at day 28 (T3/T6) when compared with baseline (T0). This will be assessed as a paired t-test comparing the mean percentage change of FIDIAL PLUS against the mean percentage change from baseline of IAL®-F at Day 28.
  Corneal endothelial cell density will be measured by non-contact specular microscopy.

SECONDARY OUTCOMES:
Incidence of a significant (≥30 mmHg) rise in IOP (Intraocular pressure) during study duration | 28 days per eye
  This will be assessed using McNemar's test to assess the difference in proportion of eyes with a significant rise in IOP during the investigation to the proportion of eyes without a significant rise in IOP during the investigation.
  IOP will be measured with Goldmann tonometer and expressed in millimeters of mercury (mmHg).
Incidence of ocular Treatment Emergent Adverse Events (TEAEs) | up to 28 days
  TEAEs are AE reported from the time of the first application of the medical device (MD).
  TEAEs will be recorded and reported on the case report form (CRF). They will be tabulated by System Organ Class (SOC) and Preferred Term (PT) after medical coding using the Medical Dictionary for Regulatory Activities (MedDRA).
Incidence of serious ocular Treatment Emergent Adverse Events | up to 28 days
  Serious TEAEs are AE reported from the time of the first application of the medical device (MD) that led to: death; to a serious deterioration in health that resulted in a life-threatening illness or injury, or resulted in a permanent impairment of a body structure or a body function, or required in-patient hospitalization or prolongation of existing hospitalization, or resulted in medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function; led to foetal distress, foetal death or a congenital abnormality or birth defect.
Change at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) of Intraocular pressure (IOP) | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  IOP will be measured with Goldmann tonometer at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) and expressed in millimeters of mercury (mmHg).
Central corneal Thickness changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  Central corneal thickness (CCT) will be measured by non-contact specular microscopy at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
Incidence and grade of anterior chamber inflammation (cells and flare measurement) | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  Assessment of anterior chamber inflammation will be performed by slit-lamp biomicroscopy at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6).
  Slit-lamp examination (SLE) will be performed before and after the instillation of dilating eye drops.
  Anterior chamber (AC) inflammation will be assessed and graded according to the SUN (Standarization of Uveitis Nomenclature) clinical scoring system.
  Anterior Chamber Cells grading:
  Grade 0, cells in field (field size is a 1 mm by 1 mm slit beam) <1 Grade 0.5+, cells in field 1-5 Grade 1+, cells in field 6-15 Grade 2+, cells in field 16-25 Grade 4+, cells in field >50
  Anterior Chamber Flare Grading:
  Grade 0, none Grade 1+, Faint Grade 2+, Moderate (iris and lens details clear) Grade 3+, Marked (iris and lens details hazy) Grade 4+, Intense (fibrin or plastic acqueous)
Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) of corneal edema | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  Epithelial corneal edema will be assessed with specular microscopy at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
Change at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) of corneal endothelial morphology | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  It will be assessed by non-contact specular microscopy at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6).
  Endothelial cell morphology will be analyzed manually or using automated measurements with the retracing method using the manufacturer's built-in image analysis software.
Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) of UDVA (Uncorrected distance visual acuity) | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  It will be measured using the Snellen chart at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6).
  Visual acuity values will be expressed in decimal, fraction or logMAR. All assessments will be performed using standard charts and procedures at specified visual angle, illumination and contrast.
Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6) of BCVA (Best corrected distance visual acuity) | Changes at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6)
  It will be measured using the Snellen chart at day 1 (T1/T4), day 7 (T2/T5) and day 28 (T3/T6).
  Visual acuity values will be expressed in decimal, fraction or logMAR. All assessments will be performed using standard charts and procedures at specified visual angle, illumination and contrast.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy